CLINICAL TRIAL: NCT04445818
Title: A Pilot Intervention Study to Increase Appreciation and Reduce Criticism Among Families in Hong Kong
Brief Title: More Appreciation and Less Criticism Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HKUSPH-MALC
Record Dates: First submitted 2020-06-16; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Parenting; Family Research; Family
Keywords: Parenting; Appreciation; Criticism; Fruit and Vegetable Consumption; Family
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Intervention Model Description: This study is a cluster randomised controlled trial with three arms: more appreciation arm (MA), less criticism arm (LC), and more fruit and vegetable arm (FV).
Masking Description: The person recruiting participants and the participants enrolled are not blinded to the allocation status. Double blinding in cluster RCTs for psychosocial or behavioural interventions is often difficult to implement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- More Appreciation (Experimental): A 6-minute engaging video will be shown, illustrating examples where a mother initially withholds her appreciation for her son's effort in school and later express it. The video will also capture the effect on the child and the family. Attributional discussion questions will follow to elicit positive outcomes of expressing appreciation and the negative outcomes of withholding appreciation (e.g., What may be the long-term effects of showing appreciation on your child, family, or on yourself?). Key points will be summarised and reinforced to enhance behavioural intention (Schwarzer & Luszczynska, 2008). Then the participants will be asked to plan by indicating when (e.g., Saturday afternoon), what (e.g., child helping a younger sibling prepare for a dictation test), and how (e.g., "I can see that you gave up your leisure time to help your sister with the spelling. Thank you!") they would express appreciation to their children.
  Interventions: Behavioral: More appreciation
- Less Criticism (Experimental): Participants will watch a 6-minute video showing examples of a father criticising his son, which will be replaced by positive communication later, and the different reactions evoked in the child and the family. Then, participants will have an attributional discussion on the negative effects of criticism (e.g., negative effect on self-worth and motivation) and positive outcomes of using constructive feedback (e.g., promptly identifying undesirable behaviours without relating to personal traits or abilities). In small groups, they will work out alternatives (i.e., constructive feedback; termed "positive reminder" in the intervention) to criticism, and each plan and write down when (e.g., after school), what (e.g., low test marks), and how (e.g., "How do you prepare for the tests?)
  Interventions: Behavioral: Less criticism
- Fruit and Vegetable (Experimental): This workshop will emphasise the importance of consuming at least 5 portions of fruit and vegetable daily for a healthy diet, and aim to boost participants' self-efficacy in achieving this. Participants will be presented with examples of one portion of fruit or vegetable, and then create their own recipes. They will also consider how to overcome obstacles of consuming more portions. Each participant will set goals and write down plans on when, where, what, and how they would increase their fruit and vegetable intake of their children and family as a whole.
  Interventions: Behavioral: More Fruit and Vegetable

INTERVENTIONS:
Behavioral: More appreciation
  Arms: More Appreciation
Behavioral: Less criticism
  Arms: Less Criticism
Behavioral: More Fruit and Vegetable
  Arms: Fruit and Vegetable

SUMMARY:
The project "More Appreciation and Less Criticism Project" (MALC) is a collaboration between the Tung Wah Group of Hospitals (TWGHs) and the School of Public Health of The University of Hong Kong (HKUSPH), funded by The Hong Kong Jockey Club Charities Trust. The objectives are to develop and test theory-driven group programmes to increase parents' intention and actual behaviours to express more appreciation or less criticism when interacting with their children, thereby enhancing family harmony and happiness.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled trial (RCT) with three arms: More Appreciation (MA), Less Criticism and Fruit and Vegetable (FV) group. Clusters, mostly schools, are the unit of random allocation to one of the three arms. Participants from all three arms will be assessed a total of four times, i.e. baseline (before the intervention workshop; (T1), immediate post-workshop (T2), 2-week post-workshop (T3) and 6-week post-workshop (T4).

"Fruit and vegetable consumption" is a subsidiary study to the More Appreciation and Less Criticism (MALC) Project. The study will take advantage of the cluster RCT design adopted by the MALC study, and aims at testing the active HAPA-based intervention (increasing fruit and vegetable intervention) delivered to the MALC control group. The fruit and vegetable group will serve as the intervention arm, and the groups that received interventions regarding increasing appreciation or decreasing criticism, served as the control arms.

ELIGIBILITY:
Inclusion Criteria:

* Parents who are Cantonese-speaking, able to complete study questionnaire, and who have children attending p.4 to p.6 will be included.

Exclusion Criteria:

* Parents with active psychiatric problems, suicidal ideations, personality disorders, emotional problems, and mental retardartion will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 803 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2013-05-31 (Actual); Study Completion 2013-05-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline self-reported appreciation behaviours at follow-ups | Baseline (before the workshop, T1), 2-week post-workshop (T3) and 6-week post-workshop (T4).
  Being assessed by averaging two items, measuring the frequency with which parents expressed appreciation (express appreciation towards children's efforts; express appreciation towards children's strengths) in the past 7 days. Responses range from 0 to 6 (0: '0 time,' 1: 'one to two times per week,' 2: 'three to four times per week,' 3: 'five to six times per week,' 4: 'once a day,' 5: 'two to three times a day,' and 6: 'four times or more per day'). The Cronbach's alpha is 0.90.
Changes from baseline self-reported criticism behaviours at follow-ups | Baseline (before the workshop, T1), 2-week post-workshop (T3) and 6-week post-workshop (T4).
  Being assessed by averaging two items, measuring the frequency with which parents expressed criticism (criticise children; express dissatisfaction towards children's behavior) in the past 7 days. Responses range from 0 to 6 (0: '0 time,' 1: 'one to two times per week,' 2: 'three to four times per week,' 3: 'five to six times per week,' 4: 'once a day,' 5: 'two to three times a day,' and 6: 'four times or more per day'). The Cronbach's alpha is 0.93.
Changes from baseline self-reported fruit and vegetable intake behaviours at follow-ups | Baseline (before the workshop, T1), 2-week post-workshop (T3) and 6-week post-workshop (T4).
  Being assessed by summing two items, one each for the number of servings of fruits and vegetables consumed in the past week.

SECONDARY OUTCOMES:
Changes from baseline outcome expectancies of more appreciation at post-workshop | Baseline (before the workshop, T1), and T2 (immediately after the workshop).
  Measured by averaging three items, "If I express my appreciation through words or action more often, my children will be more positive to themselves", "If I express my appreciation through words or action more often, my children will appreciate the other family members more", "If I express my appreciation through words or action more often, my family will be happier and more harmonious". Participants rated their agreement using a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline outcome expectancies of less criticism at post-workshop | Baseline (before the workshop, T1), and T2 (immediately after the workshop).
  Measured by averaging three items. "If I criticize my children, they will be more negative to themselves", "If I criticize my children, they will learn to criticize the other family members", "If I criticize my children, my family will be less happy and less harmonious". Participants rated their agreement using a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline outcome expectancies of fruit and vegetable intake at post-workshop | Baseline (before the workshop, T1), and T2 (immediately after the workshop).
  Measured by averaging two items. "if I eat more servings of fruit and vegetables every day, that would be good for my health", "If I eat more fruit and vegetable, I will set a good example for my children". Participants rated their agreement using a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline intention to express more appreciation at post-workshop and 2-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), and 2-week post-workshop (T3).
  Measured by a single item "In the coming 2 weeks, I intend to express appreciation to my child through words or action more often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline intention to criticize less at post-workshop and 2-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), and 2-week post-workshop (T3).
  Measured by a single item "In the coming 2 weeks, I intend to criticize my child less often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline intention of more fruit and vegetable intake at post-workshop and 2-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), and 2-week post-workshop (T3).
  Measured by a single item "in the coming 2 weeks, I intend to eat more servings of fruit and vegetables every day". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline self-efficacy of more appreciation at post-workshop and 2-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), and 2-week post-workshop (T3).
  Measured by a single item "In the coming 2 weeks, I am confident that I can express appreciation to my child through words or action more often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline self-efficacy of less criticism at post-workshop and 2-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), and 2-week post-workshop (T3).
  Measured by a single item "In the coming 2 weeks, I am confident that I can criticize my child less often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline self-efficacy of more fruit and vegetable intake at post-workshop and 2-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), and 2-week post-workshop (T3).
  Measured by a single item "In the coming 2 weeks, I am confident that I could eat more servings of fruit and vegetables every day". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline action planning of more appreciation at post-workshop, 2-week and 6-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), 2-week post-workshop (T3), and 6-week post-workshop (T4).
  Measured by a single item "In the coming 2 weeks, I have a clear plan on how to express appreciation to my child through words or action more often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline action planning of less criticism at post-workshop, 2-week and 6-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), 2-week post-workshop (T3), and 6-week post-workshop (T4).
  Measured by a single item "In the coming 2 weeks, I have a clear plan on how to criticize my child less often. Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline action planning of more fruit and vegetable intake at post-workshop, 2-week and 6-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), 2-week post-workshop (T3), and 6-week post-workshop (T4).
  Measured by a single item "In the coming 2 weeks, I have a clear plan on how to eat more servings of fruit and vegetables every day". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline coping planning of more appreciation at post-workshop, 2-week and 6-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), 2-week post-workshop (T3), and 6-week post-workshop (T4).
  Measured by a single item "In the coming 2 weeks, I have a clear plan on how to overcome challenges in expressing appreciation to my child through words or action more often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline coping planning of less criticism at post-workshop, 2-week and 6-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), 2-week post-workshop (T3), and 6-week post-workshop (T4).
  Measured by a single item "in the coming 2 weeks, I have a clear plan on how to overcome challenges to criticize my child less often". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline coping planning of more fruit and vegetable intake at post-workshop, 2-week and 6-week | Baseline (before the workshop, T1), T2 (immediately after the workshop), 2-week post-workshop (T3), and 6-week post-workshop (T4).
  Measured by a single item "In the coming 2 weeks, I have a clear plan on how to overcome challenges to eat more servings of fruit and vegetables every day". Participants rated their agreement on a 10-point scale (1 = totally disagree, 10 = totally agree).
Changes from baseline family well-being | Baseline (before the workshop, T1), 2-week post-workshop (T3) and 6-week post-workshop (T4).
  Being assessed by a composite score of 3 items, namely the 3Hs: family harmony, family happiness, and family health. Participants rated each item on a scale from 0 (not at all harmonious/ happy/ healthy) to 10 (very harmonious/ happy/ healthy). This composite score has been used in another study in Hong Kong (M. P. Wang et al., 2014) which showed a satisfactory Cronbach's alpha (0.84).

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Fung, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
Generally, individual participant data will not be shared with a third party. People not involved in the project can check the data availability from the principal investigator.

REFERENCES:
- [Result] Fung SSW, Lam TH, Sun Y, Man PKW, Ip JCM, Wan ANT, Stewart S, Ho SY. A cluster randomized controlled trial of more appreciation and less criticism in Hong Kong parents. J Fam Psychol. 2020 Sep;34(6):731-739. doi: 10.1037/fam0000628. Epub 2020 Jan 16. PMID 31944801